CLINICAL TRIAL: NCT04526327
Title: The Impact of Combination of Aerobic and Resistive Exercise on Activities of Daily Living and Risk of Fall in Osteosarcopenic Patients
Brief Title: Osteosarcopenia and Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Selda Çiftci, Principal investigator, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2189
Record Dates: First submitted 2020-08-19; First posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Sarcopenia; Osteoporosis, Osteopenia
Keywords: aerobic exercise; resistive exercise; balance; falling; physical performance; osteosarcopenia
MeSH Terms: conditions — Sarcopenia; Osteoporosis; Bone Diseases, Metabolic | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Female and male patients over 70 years of age followed-up from osteoporosis outpatient clinic
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- exercise group (Other): Female and male patients over 70 years of age with osteoporosis and sarcopenia
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — the combination of aerobic and resistive exercise, three time a week

SUMMARY:
The purpose of this study is to assess the efficacy of combination of aerobic and resistive exercise on activities of daily living and risk of fall in osteosarcopenic patients

DETAILED DESCRIPTION:
After being informed about the study and potential risk, all patients giving written informed consent will undergo study entry.

to begin with: assessment with bioelectrical body composition analyzer and first exercise and assessment clinical scales

1th month: assessment with bioelectrical body composition analyzer and assessment clinical scales 3th month: assessment with bioelectrical body composition analyzer and assessment clinical scales

ELIGIBILITY:
Inclusion Criteria:

* Over 70 years of age
* Clinical diagnosis of osteoporosis or osteopenia
* Independent mobilization
* Walking speed < 0.8 m / sec
* Grip strength < 20 kg for women, < 30 kg for men

Exclusion Criteria:

* Uncontrolled hypertension (systolic blood pressure> 200 mmHg, diastolic blood pressure> 110 mmHg)
* Uncontrolled diabetes mellitus
* Stroke, hip fracture, knee and hip arthroplasty, spinal surgery in the last 6 months
* Severe cardiac arrhythmia
* Myocardial infarction in the last 6 months
* Severe dementia and difficulties in cooperation
* Cardiac pacemaker
* Dialysis
* Acute infection
* Severe edema
* Malignancy patients
* Severe anemia (Hgb <8 mg / dl)

Ages: 70 Years to 91 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-03-03 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline on Skeletal Muscle Mass Measurement at month 3 | Baseline and Month 3
  Assessment with bioelectrical body composition analyzer male: SMI<9,2 kg/m2 female: SMI<7,4 kg/m2
Change from Baseline on Skeletal Muscle Mass Measurement at month 1 | Baseline and Month 1
  Assessment with bioelectrical body composition analyzer male: SMI<9,2 kg/m2 female: SMI<7,4 kg/m2
Change from Baseline on Katz Activities of Daily Living Scale at month 3 | Baseline and Month 3
  minimum 0, maximum 6, high scores: better
Change from Baseline on Katz Activities of Daily Living Scale at month 1 | Baseline and Month 1
  minimum 0, maximum 6, high scores: better
Change from Baseline on Short Physical Performance Battery at month 3 | Baseline and Month 3
  0-low perfomance, 12-good performance
Change from Baseline on Short Physical Performance Battery at month 1 | Baseline and Month 1
  0-low perfomance, 12-good performance
Change from Baseline on Berg Balance Test at month 3 | Baseline and Month 3
  maximum 56 point, a score of < 45 indicates individuals may be at greater risk of falling.
Change from Baseline on Berg Balance Test at month 1 | Baseline and Month 1
  maximum 56 point, a score of < 45 indicates individuals may be at greater risk of falling.
Change from Baseline on Timed Up and Go Test at month 3 | Baseline and Month 3
  Stand up and walk 3 meters, turn around, walks back to the chair and sit down.14 seconds or longer : high risk for falling
Change from Baseline on Timed Up and Go Test at month 1 | Baseline and Month 1
  Stand up and walk 3 meters, turn around, walks back to the chair and sit down.14 seconds or longer : high risk for falling
Change from Baseline on Five Times Sit to Stand Test at month 3 | Baseline and Month 3
  Lower times: better scores
Change from Baseline on Five Times Sit to Stand Test at month 1 | Baseline and Month 1
  Lower times: better scores

CONTACTS AND LOCATIONS:
Overall Officials: Figen Yılmaz, Study Chair — Şişli Hamidiye Etfal Training and Research Hospital
Locations (1):
- Şişli Hamidiye Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No